CLINICAL TRIAL: NCT06207604
Title: Survivability of Dental Implants Placed in Atrophic Maxillae Using Open Sinus Elevation Technique With and Without Bone Grafting Material. A Randomized Controlled Clinical Trial
Brief Title: Implant Placement Using Open Sinus Elevation Technique With and Without Bone Grafting Material
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Clinical director of implant speciality program, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDCE.N8
Record Dates: First submitted 2023-12-17; First posted 2024-01-17 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Sinus Elevation
Keywords: dental implants; bone grafting; posterior maxilla
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open sinus lifting without bone grafting and simultaneous implant placement (Experimental): When adequate release of the membrane is achieved and deemed enough by the operator, an osteotomy is created in the edentulous area following the drilling sequence provided by the implant system used. the implant placement is done directly with the implant motor and the use of a hand driver if needed to adjust the implant platform relation to the crestal bone, followed by cover screw placement.
  Interventions: Procedure: Open sinus lifting without bone grafting and simultaneous implant placement
- Open sinus lifting with bone grafting and simultaneous implant placement (Active Comparator): When adequate release of the membrane is achieved and deemed enough by the operator, an osteotomy is created in the edentulous area following the drilling sequence provided by the implant system used. the palatal packing of bone is made before the implant placement, as the palatal aspect of the sinus will be inaccessible after placement of the implant, the implant placement is done directly with the implant motor and the use of a hand driver if needed to adjust the implant platform relation to the crestal bone, followed by cover screw placement.
  Interventions: Procedure: Open sinus lifting with bone grafting and simultaneous implant placement

INTERVENTIONS:
Procedure: Open sinus lifting without bone grafting and simultaneous implant placement — no bone graft will be used after open sinus lifting
  Arms: Open sinus lifting without bone grafting and simultaneous implant placement
Procedure: Open sinus lifting with bone grafting and simultaneous implant placement — bone graft will be packed palatally after open sinus elevation and before implant placement, then implant placement will took place followed by packing of bone grafts
  Arms: Open sinus lifting with bone grafting and simultaneous implant placement

SUMMARY:
The success rate of dental implants after graftless sinus augmentation versus conventional sinus augmentation surgery in atrophic maxillae in edentulous patients was investigated and it was concluded that despite the bone gain in ten garftless side, implant survival were significantly lower in the non-grafted side. One year later, Lie et al., conducted a systematic review to evaluate efficacy of graftless maxillary sinus membrane elevation using the lateral window approach for implantation in the atrophic maxilla. It showed a high implant survival rate in non-grafted maxillary sinus lifts and conventional sinus lifts using augmentation materials and there was no significant difference in the ISQ values between both procedures. However, further randomized clinical trials with long-term follow-up were recommended.

DETAILED DESCRIPTION:
It is well documented in literature that after dental extractions, the alveolar ridge will undergo some changes in volume both in hard and soft tissue both in the anterior and posterior region of the oral cavity. This adds challenges to properly place dental implants following tooth extraction in a good prosthetic position, specifically in the Maxillary posterior region due to the proximity of the Maxillary Sinus. Maxillary sinus pneumatization is an ongoing process that occurs naturally causing increased maxillary sinus volume on the expense of the alveolar ridge. When the combination of sinus pneumatization and bony atrophy of the maxilla occurs following tooth extractions together over time, the edentulous ridge dimension can be very minimal.

Numerous techniques were suggested to facilitate implant placement in atrophic posterior maxilla. The first proposed technique was the Maxillary Open sinus technique, it was first proposed by Dr. O. Hilt Tatum at an implant meeting in Alabama, however, Boyne and James in 1980 were the first to publish this surgical technique. In order to regain the vertical dimension, open sinus technique was originally performed in a staged manner over two steps, where the implant was placed after a healing period after Maxillary sinus augmentation, however, the different sinus elevation techniques, whether staged or one step did not seem to affect the implant success rate and showed bone gain of up to 12 mm.

Some authors suggested less invasive techniques that were of less discomfort to the patient, more cost effective and less time consuming. Summers proposed the osteotome technique, where similar to traditional drilling, an osteotomy is prepared using a set of osteotomes 1mm short of the sinus floor, followed by fracturing of the floor using the proper sized osteotome with bone graft material, which will allow the introduction of bone grafting material into the sinus floor, followed by the placement of the dental implant. However it was limited to 5 mm in terms of bone gain compared to 12 mm bone gain in the open sinus technique. Over the years, modifications to Summers original technique were made. Short dental implants were proposed; however, a review of the literature reveals implants shorter than 10 mm often have a higher failure rate than longer implants. These complications may be related to an increase in crown height, higher bite forces in the posterior regions, and less bone density. As a result, methods to decrease stresses to the bone-implant interface are to be researched. This necessitates and puts the clinician in a situation where the open sinus procedure is sometimes inevitable.

The formation of bone in elevated sinus space was a mystery and its reason was unknown. However a histological study showed the osteogenic potential of the Schneiderian membrane when it was subcutaneously placed in rats suggesting that bone genesis could be directly related to the presence of the Schneiderian membrane in the maxillary sinus regardless the presence or absence of a bone grafting material. This technique was based on the concept that the lifting of the sinus membrane and the establishment of a compartment with a blood clot could result in new bone around the inserted implants in a similar way that bone-graft materials maintain the augmented space and promote osteogenesis.

ELIGIBILITY:
Inclusion Criteria:

1. Edentulous atrophic posterior maxillary ridge.
2. Residual alveolar ridge height within 3-5mm.
3. At least 2mm band of keratinized tissue.
4. Patients with good oral hygiene.
5. Compliant patients to the follow up periods.

Exclusion Criteria:

1. Medically compromised patients.
2. Smokers.
3. Pregnant females.
4. Patients with active periodontal disease.
5. Bruxer patients.
6. Patients with chronic or active sinusitis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Long- term Implant Stability | 12 months
  Resonance frequency analysis will be employed with a dedicated device (Osstell).

SECONDARY OUTCOMES:
Implant survivability | 12 months
  Individual unattached implant that is immobile when tested clinically, radiography that does not demonstrate evidence of peri-implant radiolucency, Bone loss that is less than 0.2 mm annually after the implant's first year of service, No persistent pain, discomfort or infection
Vertical bone height formed | 12 months
  CBCTS

IPD SHARING:
Plan to Share IPD: No